CLINICAL TRIAL: NCT01033916
Title: Strict or Liberal Insulin Protocol Following Coronary Artery Bypass Graft (CABG) Surgery
Acronym: SLIP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inova Health Care Services (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SLIP - 09.111
Record Dates: First submitted 2009-12-16; First posted 2009-12-17 (Estimated); Last update posted 2022-01-06 (Actual); Status verified 2022-01

CONDITIONS: Blood Glucose; Coronary Artery Bypass; Insulin; Coronary Disease
Keywords: Blood Glucose; Insulin/Administration and Dosage; Coronary Artery Bypass
MeSH Terms: conditions — Insulin Resistance; Coronary Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- STRICT Glucose Control (80-120 mg/dL) (No Intervention): The STRICT arm of the study will have a target Blood Glucose level ranging from 80-120 mg/dL. This is currently the standard of care for post CABG patients.
- LIBERAL (Target Glucose:121-180 mg/dL) (Active Comparator)
  Interventions: Other: LIBERAL

INTERVENTIONS:
Other: LIBERAL — The LIBERAL arm of the study will have a target Blood Glucose level ranging from 121-180 mg/dL. As opposed to the standard of less than 120 mg/dL.
  Arms: LIBERAL (Target Glucose:121-180 mg/dL)

SUMMARY:
This research study is designed to better understand post-operative complications as related to the tightness of blood sugar control. It is also hoped that we may learn that a more liberal control of your blood sugars is not inferior to the current strict glucose control. Our ultimate goal is to evaluate if there is any change in the rates of complications between the two groups. We will be comparing the current strict blood glucose control with a more liberal target for blood sugars.

DETAILED DESCRIPTION:
Hyperglycemia is commonly encountered following cardiac surgery, whether a patient has a history of diabetes or not. Hyperglycemia has been associated with increased perioperative morbidity and mortality; several studies have demonstrated that glycemic control utilizing insulin protocols improves operative mortality, lowers operative morbidity (mediastinitis, atrial fibrillation), and improves long-term survival. However, the optimal target for serum glucose has not been established in post-CABG patients.

Methods:

All CABG patients will be consented prior to surgery. Inclusion criteria for non-diabetic patient is a random fingerstick blood glucose (FSBG) above >150 mg/dL prior, during, or immediately following surgery. All patients with history of diabetes mellitus (Type 1 or Type II) will be immediately eligible for inclusion.

Following CABG surgery, if the patient was started intra-operatively on an insulin infusion, then that patient will be randomized to one of two treatment target groups: Group 1 [Blood Glucose (BG): 80 mg/dL-120 mg/dL] or Group 2 [BG: 121-180 mg/dL]. The randomization design will be a 1:1 allocation of patients between the two groups, with both diabetic and non-diabetic patients enrolled in both arms of the study. Patients will be maintained on an electronic-based protocol of intravenous insulin for a minimum of 72 hrs postoperatively. Patients remaining in the CVICU greater than 72 hrs will have their intravenous insulin continued until transfer to the step-down unit.

The Glucommander© will be programmed to adjust the insulin drip to one of these two target groups. The nursing staff will not be blinded to treatment group allocation. The primary endpoint with be a composite of operative death, major adverse cardiac events (MACE: death, myocardial infarction, re-vascularization), STS Defined Major Morbidity (re-operation, Cerebrovascular accident, Deep Sternal Wound Infection/Mediastinitis, Prolonged Ventilatory Support (> 24 hrs), Acute Renal Failure), and prolonged inotropic support. The pre-specified sub-group analysis will compare perioperative outcome of patients with diabetes vs non-diabetic patients.

Hypothesis:

Our hypothesis is that the perioperative outcome of Group 2 [BG: 121 - 180 mg/dL] will not be inferior to Group 1 [BG: 80-120 mg/dL]. We anticipate significantly more hypoglycemic events in Group 1.

ELIGIBILITY:
Inclusion Criteria:

1. All diabetic patients going for isolated, non-emergent CABG surgery at Inova Fairfax Hospital (IFH).
2. Non diabetic patients going for isolated, non-emergent CABG Surgery at IFH that are found to have a finger stick blood glucose > 150 mg/dl, either pre-operative, during the procedure or post-operatively.
3. Those patients that meet Inclusion Criteria #1 OR #2 AND have been started on an insulin infusion while in the operative room will be enrolled.

Exclusion Criteria:

1. Patients that are not undergoing CABG surgery.
2. Patients that post-CABG surgery are not on an insulin infusion.
3. Patients that are undergoing other procedures in addition to CABG will be excluded. (ie. CABG + valve repair)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2009-12-01 (Actual); Primary Completion 2011-04-30 (Actual); Study Completion 2016-07-30 (Actual)

PRIMARY OUTCOMES:
Operative death, major adverse cardiac events (death, myocardial infarction, re-vascularization), re-operation, Cerebrovascular accident, Deep Sternal Wound Infection, Prolonged Ventilatory Support, Acute Renal Failure, and prolonged inotropic support. | 30 days

SECONDARY OUTCOMES:
The second pre-specified endpoint will be all-cause mortality at 90 days. | 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Niv Ad, MD, Principal Investigator — Inova Heart & Vascular Institute
Locations (1):
- Inova Fairfax Hospital, Falls Church, Virginia, United States